CLINICAL TRIAL: NCT00122759
Title: Prospective Study on the Cost-Effectiveness of Adding Ketamine to Midazolam-Sufentanil Sedation Regimen in Mechanically Ventilated Patients
Brief Title: Ketamine Sedation in Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMR3
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Respiratory Insufficiency; Pain; Psychomotor Agitation
Keywords: Mechanical ventilation; Agitation
MeSH Terms: conditions — Respiratory Insufficiency; Pain; Psychomotor Agitation | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ketamine

SUMMARY:
* Adequate sedation is of paramount importance to avoid stress and pain in mechanically ventilated patients. It is usually achieved by infusing sedatives (benzodiazepine) and analgesic (opiate) drugs.
* This combined sedation may not be sufficient in some instances.
* The aim of this study is to evaluate whether addition of a third substance, ketamine, allows the achievement of better sedation and avoids the use of neuromuscular blocking agents.

DETAILED DESCRIPTION:
* Mechanical ventilation is widely used in critically ill patients. Sedation is used in most instances to alleviate symptoms of pain and distress. It usually consists of an association of opiates and benzodiazepines.
* In some instances, pain and agitation persist despite this combined sedation regimen. In such cases, the clinicians have the choice between increasing dosage of these 2 substances which may increase their adverse effects (mainly hypotension) and/or adding a neuromuscular blocking agent which is not devoid of adverse effects (mainly the onset of neuromyopathy of critical illness).
* This study will assess the safety, efficacy and cost-effectiveness of adding ketamine, a well known anesthetic agent, to a combination of midazolam and sufentanil when this combination is not sufficient to reach acceptable sedation target.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients who receive adequate dosing of sedative agents (midazolam > 0.15 mg/kg/h plus sufentanil > 0.3 mcg/kg/h)
* Persistence of agitation indicating that sedation is not appropriate, as assessed by validated sedation scales (Harris scare; Motor Activity Assessment scale).

Exclusion Criteria:

* Pregnancy
* Patient who already receives neuromuscular blocking agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-12; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of the adequacy of sedation in patients receiving benzodiazepine plus opiate or this combination plus adjunctive ketamine
Comparison of the cost of sedation with both regimens

SECONDARY OUTCOMES:
Overall duration of mechanical ventilation
Need to administer neuromuscular blocking agents

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Réanimation Médicale, Hôpital Louis Mourier, Colombes, France

REFERENCES:
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Ostermann ME, Keenan SP, Seiferling RA, Sibbald WJ. Sedation in the intensive care unit: a systematic review. JAMA. 2000 Mar 15;283(11):1451-9. doi: 10.1001/jama.283.11.1451. PMID 10732935
- [Background] Bourgoin A, Albanese J, Leone M, Sampol-Manos E, Viviand X, Martin C. Effects of sufentanil or ketamine administered in target-controlled infusion on the cerebral hemodynamics of severely brain-injured patients. Crit Care Med. 2005 May;33(5):1109-13. doi: 10.1097/01.ccm.0000162491.26292.98. PMID 15891344